CLINICAL TRIAL: NCT06535529
Title: Acetazolamide Versus Dapagliflozin in Acute Decompensated Heart Failure Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mahmoud I Mostafa, Lecturer of Clinical Pharmacy.Lecturer of Clinical Pharmacy, Faculty of Pharmacy, Helwan University, Cairo, Egypt., Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acetazolamide vs Dapa in ADHF
Record Dates: First submitted 2024-06-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute Heart failure; ADHF; Acetazolamide; SGLT2 inhibitors; SGLT2i
MeSH Terms: interventions — Acetazolamide; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, randomized, two-armed parallel comparator study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide + Standard Care (Active Comparator): Participants in this arm will receive:
  1. Acetazolamide: 500 mg orally, once daily for 3 days
  2. Intravenous loop diuretics: Administered at double the oral maintenance dose, given as follows:
     * Initial dose: Single bolus immediately after randomization
     * Subsequent doses: Split into two or more doses (separated by ≥6 hours) on each of the next 2 days The specific loop diuretic used (e.g., furosemide) will be determined by the treating physician based on the patient's prior medication regimen and clinical status.
  Interventions: Drug: Acetazolamide
- Dapagliflozin + Standard Care (Active Comparator): Participants in this arm will receive:
  1. Dapagliflozin: 10 mg orally, once daily for 3 days
  2. Intravenous loop diuretics: Administered as described in Arm 1
  Interventions: Drug: Dapagliflozin 10mg

INTERVENTIONS:
Drug: Acetazolamide — Patients will receive acetazolamide 500 mg once daily for 3 days as add on therapy to IV loop diuretics
  Other Names: Cidamix
  Arms: Acetazolamide + Standard Care
Drug: Dapagliflozin 10mg — patient will receive oral dapagliflozin 10 mg once daily for 3 days as add on therapy to IV loop diuretics
  Other Names: Forxiga
  Arms: Dapagliflozin + Standard Care

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of acetazolamide versus dapagliflozin as an add-on in treating acute decompensated heart failure (ADHF) in adult patients with clinical signs of volume overload requiring intravenous loop diuretics. It will also assess the safety of these drugs when added to standard care. The main questions it aims to answer are:

* Does acetazolamide or dapagliflozin lead to a greater reduction in N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels?
* Which drug results in better loop diuretic efficiency, as measured by weight loss per 40 mg of intravenous furosemide or equivalent? We will compare acetazolamide to dapagliflozin, both added to standard intravenous loop diuretic therapy, to see which is more effective in decongesting patients with ADHF.

Participants will:

* Take either acetazolamide or dapagliflozin orally every day for 3 days
* Receive intravenous loop diuretics as part of standard care
* Undergo regular assessments of heart failure symptoms, weight, and laboratory tests
* Be followed up until hospital discharge and for 30 days after starting the study

DETAILED DESCRIPTION:
A. Study design

* Prospective, open-label, randomized, two-armed parallel comparator study.
* Participants recruited in the study must provide written informed consent after obtaining ethical approval from ethics committee.

B. Study settings Critical Care Medicine Department - Cairo University Hospitals. C. Population of study Adult patients who are admitted to Critical Care Medicine Department - Cairo University Hospitals because of acute decompensated heart failure will be screened for inclusion into the study. Patients who have at least one clinical sign of volume overload (i.e., edema, pleural effusion, or ascites) and ECHO-confirmed HF at screening will be included in the study.

D.Treatment :

I.V loop diuretics

At the moment of randomization, oral loop diuretics are stopped. Patients need to empty their bladder before administration of the first dose of loop diuretics and all will receive an intravenous loop diuretic at double the oral maintenance dose, administered as a single bolus immediately after randomization and split into more than two doses (separated by ≥6 hours) on each of the next 2 days.

Group 1: Oral Acetazolamide Together with the initial bolus dose of loop diuretics, patients will receive 500 mg oral Acetazolamide. Time of subsequent dose of acetazolamide taken once daily will start together with the first maintenance loop diuretic dose.

Group 2: Oral Dapagliflozin Together with the initial dose of loop diuretics, patients will receive 10 mg Dapagliflozin.

Time of subsequent dose of Dapagliflozin taken once daily will start together with the first maintenance loop diuretic dose.

E. Study tools

Modified ADVOR Score The modified ADVOR congestion score will be calculated on a scale from 0 to 10 based on the sum of scores for the degree of edema (0 to 4), pleural effusion (0 to 3), and ascites (0 to 3), with higher scores indicating a worse condition on all scales. This score will be calculated for each included patient before the administration of the first dose of diuretics during the treatment phase, at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of 18 years of age or older.
* An elective or emergency hospital admission with clinical diagnosis of decompensated HF with at least one clinical sign of volume overload (e.g. edema, ascites confirmed by echography or pleural effusion confirmed by chest X-ray or echography).
* Assessed LVEF by any imaging technique; i.e. echocardiography, catheterization, nuclear scan magnetic resonance imaging within 12 months of inclusion.

Exclusion Criteria:

* The receipt of acetazolamide maintenance therapy.
* Receipt of an SGLT2 inhibitor in the 48 hours before randomization.
* An estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2.
* Use of any non-protocol defined diuretic agent with the exception of mineralocorticoid receptor antagonists during the treatment phase of the study. Thiazides, metolazone, indapamide and amiloride should be stopped upon study inclusion. If patient is taking a combination drug including a thiazide-type diuretic, the thiazide-type diuretic should be stopped.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-24 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | From baseline to day 5 or intensive care unit (ICU) discharge, whichever occurs first
  Absolute change in NT-proBNP levels from baseline to end of study period
calculating of weight loss Loop diuretic efficiency | 72 hours from initiation of treatment
  Weight loss (in kg) per 40 mg of intravenous furosemide or equivalent dose of other loop diuretics

SECONDARY OUTCOMES:
Number of Participants with Successful decongestion | 72 hours from initiation of treatment
  Proportion of patients achieving an ADVOR Score ≤ 1 without the need for escalating diuretic strategy (defined as doubling loop diuretic dose, addition of chlorthalidone, or ultrafiltration)
Duration of the index hospital admission | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 100 weeks
  Number of days from randomization until the date of discharge
30-day mortality | Up to 30 days
  Proportion of patients who die from any cause within 30 days of randomization
Cumulative dose of intravenous loop diuretics | 5 days
  Total milligrams of intravenous furosemide or equivalent dose of other loop diuretics administered
Incidence of treatment-related metabolic acidosis | 5 days
  Proportion of patients developing metabolic acidosis requiring sodium bicarbonate (NaHCO3) supplementation
percent of worsening renal failure (WRF) | up to 4 weeks
  Proportion of patients experiencing either: a) An increase in serum creatinine > 0.3 mg/dL from baseline, or b) A decrease in estimated glomerular filtration rate (eGFR) > 20% from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Critical Care Medicine Department - Cairo University Hospitals., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mullens W, Verbrugge FH, Nijst P, Martens P, Tartaglia K, Theunissen E, Bruckers L, Droogne W, Troisfontaines P, Damman K, Lassus J, Mebazaa A, Filippatos G, Ruschitzka F, Dupont M. Rationale and design of the ADVOR (Acetazolamide in Decompensated Heart Failure with Volume Overload) trial. Eur J Heart Fail. 2018 Nov;20(11):1591-1600. doi: 10.1002/ejhf.1307. Epub 2018 Sep 21. PMID 30238574
- [Background] Mullens W, Dauw J, Martens P, Verbrugge FH, Nijst P, Meekers E, Tartaglia K, Chenot F, Moubayed S, Dierckx R, Blouard P, Troisfontaines P, Derthoo D, Smolders W, Bruckers L, Droogne W, Ter Maaten JM, Damman K, Lassus J, Mebazaa A, Filippatos G, Ruschitzka F, Dupont M; ADVOR Study Group. Acetazolamide in Acute Decompensated Heart Failure with Volume Overload. N Engl J Med. 2022 Sep 29;387(13):1185-1195. doi: 10.1056/NEJMoa2203094. Epub 2022 Aug 27. PMID 36027559
- [Background] Mullens W, Schulze PC, Westphal J, Bogoviku J, Bauersachs J. Great debate: in patients with decompensated heart failure, acetazolamide in addition to loop diuretics is the first choice. Eur Heart J. 2023 Jun 25;44(24):2159-2169. doi: 10.1093/eurheartj/ehad266. PMID 37207453
- [Background] Malik BA, Nnodebe I, Fayaz A, Inayat H, Murtaza SF, Umer M, Zaidi SAT, Amin A. Effect of Acetazolamide as Add-On Diuretic Therapy in Patients With Heart Failure: A Meta-Analysis. Cureus. 2023 Apr 18;15(4):e37792. doi: 10.7759/cureus.37792. eCollection 2023 Apr. PMID 37213994
- [Background] Sabina M, Barakat Z, Feliciano A, Lamb A, Alsamman MM. Unlocking the Potential of Acetazolamide: A Literature Review of an Adjunctive Approach in Heart Failure Management. J Clin Med. 2024 Jan 4;13(1):288. doi: 10.3390/jcm13010288. PMID 38202295
- [Background] Kosiorek A, Urban S, Detyna J, Biegus J, Hurkacz M, Zymlinski R. Diuretic, natriuretic, and chloride-regaining effects of oral acetazolamide as an add-on therapy for acute heart failure with volume overload: a single-center, prospective, randomized study. Pol Arch Intern Med. 2023 Dec 21;133(12):16526. doi: 10.20452/pamw.16526. Epub 2023 Jul 6. PMID 37415505
- [Background] Siddiqi AK, Maniya MT, Alam MT, Ambrosy AP, Fudim M, Greene SJ, Khan MS. Acetazolamide as an Adjunctive Diuretic Therapy for Patients with Acute Decompensated Heart Failure: A Systematic Review and Meta-Analysis. Am J Cardiovasc Drugs. 2024 Mar;24(2):273-284. doi: 10.1007/s40256-024-00633-9. Epub 2024 Feb 28. PMID 38416359
- [Background] Cox ZL, Collins SP, Hernandez GA, McRae AT 3rd, Davidson BT, Adams K, Aaron M, Cunningham L, Jenkins CA, Lindsell CJ, Harrell FE Jr, Kampe C, Miller KF, Stubblefield WB, Lindenfeld J. Efficacy and Safety of Dapagliflozin in Patients With Acute Heart Failure. J Am Coll Cardiol. 2024 Apr 9;83(14):1295-1306. doi: 10.1016/j.jacc.2024.02.009. PMID 38569758